CLINICAL TRIAL: NCT04068922
Title: Adaptability and Resilience in Aging Adults-2
Acronym: ARIAA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802729; 5R00AG052642-05 (NIH); 5K99AG052642-02 (NIH)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Aging; Chronic Low-back Pain
Keywords: aging; resilience; low back pain; positive affect; hope; self-efficacy; acceptance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilience Intervention (Experimental): Participants will initially complete a baseline assessment assessing study eligibility. The Resilience intervention consists of seven weekly 1.5-hour group sessions guided by trained clinicians. Due to the COVID-19 pandemic, these group session may be conducted through Zoom. Skills and content will be directed toward improving pain management by enhancing positive emotions, setting goals, learning to live a life according to one's values, and boosting self-confidence in one's ability to manage pain. Self-administered activities include the identification of personal strengths, pleasant activity scheduling, expressing gratitude, values clarification, mindfulness practice, goal setting, positive reappraisal, and noting positive events.
  Interventions: Behavioral: Resilience Intervention

INTERVENTIONS:
Behavioral: Resilience Intervention — Resilience skills training including: pleasant activities, hope/goal-setting, pain acceptance, positive events/reappraisals, and self-efficacy.

SUMMARY:
Chronic low back pain is a major health concern among older adults and is associated with increased economic, functional, and psychological burden. Resilience has been highlighted as a crucial factor in positive health-related functioning, and a growing body of literature supports the use of resilience-based interventions in chronic pain. Therefore, the goals of this project are to examine the feasibility and acceptability of a resilience intervention for chronic low back pain among older adults.

DETAILED DESCRIPTION:
Chronic pain is one of the leading causes of disability, affecting over 100 million people in the United States and resulting in tremendous health care costs and psychological burden. Older adults are disproportionately impacted by pain, with an estimated 60-70% of people over the age of 65 reporting persistent pain. Despite this, pain management is frequently suboptimal among older adults as pharmacological therapies show limited clinical efficacy and a greater risk of adverse effects, and nonpharmacological (e.g., psychological) treatments are often underutilized.

Resilience is conceptualized as adaptive functioning in the face of adversity and comprises a range of psychological, social, and physical resources. Increasing evidence suggests that modifiable resilience factors are associated with more favorable pain outcomes, including lower clinical pain/disability, higher quality of life, and enhanced psychological and physical functioning. Although cross-sectional research supports the significance of these resilience factors in pain adaptation, and positive psychological therapies have been shown to yield improvements in health and well-being, strategies to augment resilience are understudied in individuals with chronic pain.

Using a Stage Model approach,the aim of this project is to conduct a Stage I pilot study and examine the feasibility and acceptability of a resilience intervention for chronic low back pain among older adults. Intervention modules will specifically engage hope, self-efficacy, positive affect, and pain acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Low back pain on at least half the days over the previous 6 months
* Average daily back pain score ≥3 on a 0-10 numerical rating scale
* At least moderate (≥3/10) CLBP-related interference on a 0-10 numerical rating scale
* Able to read/write in English

Exclusion Criteria:

* Current participation in another psychological treatment
* Severe psychiatric illness not adequately controlled by medication (e.g., schizophrenia, bipolar disorder) or other conditions anticipated to impair intervention engagement (e.g., substance abuse/dependence)
* Presence of chronic, malignant pain (e.g., HIV, cancer) or systemic inflammatory disease (e.g., rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, etc.)
* Significant cognitive impairment on the MoCA
* If currently taking prescription analgesic or psychotropic medication, must be stabilized on these treatments for ≥4 weeks prior to the baseline assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Bartley, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lysne PE, Palit S, Morais CA, DeMonte LC, Lakdawala M, Sibille KT, Bartley EJ. Adaptability and Resilience in Aging Adults (ARIAA): protocol for a pilot and feasibility study in chronic low back pain. Pilot Feasibility Stud. 2021 Oct 19;7(1):188. doi: 10.1186/s40814-021-00923-y. PMID 34666839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this single-arm clinical trial began in January 2020, with the last participant enrolled in July 2022. Participants with chronic low back pain were recruited via provider referral, study flyers, radio and newspaper advertisement, health fairs, social media, and registries maintained by the Pain Research & Intervention Center of Excellence and the Clinical and Translational Science Institute at the University of Florida.
Pre-assignment Details: Of the 200 individuals who expressed interest in the study or who met initial eligibility criteria, 63 participants were eligible and enrolled. Of the 63 individuals who were enrolled, 94% of participants commenced treatment.
Groups:
- Resilience Intervention: The Resilience intervention consisted of seven weekly 1.5-hour group sessions guided by trained clinicians. Skills and content targeted positive emotions, setting goals, learning to live a life according to one's values, and boosting self-confidence in one's ability to manage pain. Self-administered activities included the identification of personal strengths, pleasant activity scheduling, expressing gratitude, values clarification, mindfulness practice, goal setting, positive reappraisal, and noting positive events.
  Resilience Intervention: Resilience skills training including: pleasant activities, hope/goal-setting, pain acceptance, positive events/reappraisals, and self-efficacy.
Period: Overall Study
Arm/Group | Resilience Intervention
Started | 63 (63 participants were eligible and enrolled.)
Received Intervention | 59
Completed | 50
Not Completed | 13
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Number represents the participants who completed the intervention (out of 59 who were enrolled and commenced the intervention)
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.98 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Session-level Engagement
Description: Treatment Engagement Questionnaire: 6-item study-adapted questionnaire assessing perceptions of engagement, interest in the session content, and usefulness of the home activities. Items are rated on a 0 to 8 scale and mean scored, with the mean value across sessions calculated. Higher scores indicate greater treatment engagement.
Time Frame: Assessed Weekly up to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
score on a scale | 6.3 (1.0)

2. Primary Outcome: Treatment Satisfaction
Description: 8-item Client Satisfaction Questionnaire: Response to self-reported quality of the treatment, willingness to recommend the treatment, and general satisfaction with the treatment. Items are rated on a 1 to 4 scale with the mean value calculated. Higher scores indicate greater satisfaction with the treatment.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
score on a scale | 3.4 (0.50)

3. Primary Outcome: Treatment Credibility and Expectancy
Description: Treatment Expectation Questionnaire: 7-item study-adapted questionnaire assessing the credibility and reasonableness of the intervention, and expectation for change in pain symptoms. Items are rated on a 0 to 10 scale. A mean score is calculated for the questionnaire, with higher scores indicating greater treatment credibility.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
score on a scale | 7.7 (1.6)

4. Primary Outcome: Satisfaction With Intervention Content
Description: Intervention Content Satisfaction Questionnaire: 33-item study-developed questionnaire assessing the usefulness of each intervention session module and home activity. Items are rated on a 0 to 4 scale with the mean value calculated. Higher scores indicate greater satisfaction with the intervention content.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
score on a scale | 2.9 (0.78)

5. Primary Outcome: Intervention Commencement Rate
Description: Percentage of participants who are enrolled in the study and commence treatment/intervention.
Time Frame: Baseline to Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 63
Participants | 59

6. Primary Outcome: Participant Retention
Description: Percentage of participants who commence treatment/intervention and complete the 8-week time-point.
Time Frame: Baseline to 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 59
Participants | 50

7. Primary Outcome: Questionnaire Feasibility
Description: Percentage completion rates of primary outcome study measures (averaged across all sessions).
Time Frame: Baseline to 8 Weeks
Measure: Mean (Full Range); unit: percentage of completion
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
percentage of completion | 96.8 [92.0 to 100.0]

8. Primary Outcome: Home Activity Feasibility
Description: Home Activities Questionnaire: 3-item study-adapted questionnaire assessing the degree of home-activity completion, level of understanding regarding home activities, and degree of time and effort needed to complete activities. Items are rated on a 0 to 6 scale and mean scored, with the mean value across sessions calculated. Higher scores indicate greater feasibility of home activity completion.
Time Frame: Assessed Weekly up to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resilience Intervention
Number analyzed (Participants) | 50
score on a scale | 4.6 (0.88)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Resilience Intervention
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 8/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resilience Intervention (N=63)
Bladder Infection (Renal and urinary disorders) | 1
Fractured Toe (Musculoskeletal and connective tissue disorders) | 1
Blood Clot (Blood and lymphatic system disorders) | 1
Enlarged Prostate (Reproductive system and breast disorders) | 1
Severe Back Pain and Numbness in Leg (Musculoskeletal and connective tissue disorders) | 1
Heart Attack (Cardiac disorders) | 1
Unspecified Illness (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04068922/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT04068922/ICF_001.pdf